CLINICAL TRIAL: NCT00164736
Title: HIV Infection and Breastfeeding: Interventions for Maternal and Infant Health
Brief Title: Breastfeeding, Antiretroviral, and Nutrition Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina, Chapel Hill (Other); Kamuzu Central Hospital (Other)
Responsible Party: Dr. Denise Jamieson, CDC
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-3946; U48CCU409660 (Other Grant/Funding Number: U.S. Centers for Disease Control and Prevention); PA 04003 SIP 26-04 (Other Grant/Funding Number: U.S. Centers for Disease Control and Prevention)
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infections
Keywords: HIV; Clinical trial; breastfeeding; mother-to-child-transmission; nutrition; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Zidovudine; Lamivudine; Lopinavir; Ritonavir; Nevirapine; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Maternal ARVs & Nutrition Supplement (Active Comparator): Extended maternal ARVs for prophylaxis (for the infant) & daily nutritional supplement given to the mother
  Interventions: Drug: Maternal zidovudine/lamivudine/lopinavir-ritonavir; Dietary Supplement: Maternal protein and calorie supplement
- Infant NVP & Nutrition Supplement (Active Comparator): Extended infant nevirapine for prophylaxis & daily nutritional supplment given to the mother
  Interventions: Drug: Infant nevirapine; Dietary Supplement: Maternal protein and calorie supplement
- Maternal ARVs & No Nutrition Supplement (Active Comparator): Extended maternal ARVs for prophylaxis (for the infant) & no nutritional supplement given to the mother
  Interventions: Drug: Maternal zidovudine/lamivudine/lopinavir-ritonavir
- Infant NVP & No Nutrition Supplement (Active Comparator): Extended infant nevirapine for prophylaxis & no nutritional supplment given to the mother
  Interventions: Drug: Infant nevirapine
- No Drugs & Nutrition Supplement (Active Comparator): No extended maternal ARV prophylaxis nor infant nevirapine prophylaxis & daily nutritional supplement given to the mother.
  Note: As of March 2008, the third arm of the antiretroviral intervention, in which neither mother nor infant received drugs beyond enhanced standard of care, was stopped based on recommendations of a Data and Safety Monitoring Board review of interim efficacy results and safety data after 77% participants had received treatment assignment.
  Interventions: Dietary Supplement: Maternal protein and calorie supplement
- No Drugs & No Nutrition Supplement (No Intervention): No extended maternal ARV prophylaxis nor infant nevirapine prophylaxis & no nutritional supplement given to the mother.
  Note: As of March 2008, the third arm of the antiretroviral intervention, in which neither mother nor infant received drugs beyond enhanced standard of care, was stopped based on recommendations of a Data and Safety Monitoring Board review of interim efficacy results and safety data after 77% participants had received treatment assignment.

INTERVENTIONS:
Drug: Maternal zidovudine/lamivudine/lopinavir-ritonavir — Total daily dose: zidovudine 600mg, lamivudine 300mg, (taken as Combivir 1 tab twice a day with food). Lopinavir/ritonavir 400/100mg (taken as 2 tabs twice a day). Commencing after delivery and through to 28 weeks.
  Other Names: Combivir tabs (zidovudine 300mg and lamivudine 150mg); Aluvia tabs (lopinavir 200mg /ritonavir 50mg)
  Arms: Maternal ARVs & No Nutrition Supplement; Maternal ARVs & Nutrition Supplement
Drug: Infant nevirapine — Nevirapine suspension once daily dose. 0-14days: 10mg; 3-18weeks: 20mg; 19-28weeks: 30mg.
  To 28 weeks while breastfeeding.
  Other Names: Viramune (Nevirapine) suspension 50mg/5ml
  Arms: Infant NVP & No Nutrition Supplement; Infant NVP & Nutrition Supplement
Dietary Supplement: Maternal protein and calorie supplement — High energy, nutrient-dense, micronutrient fortified nutritional supplement. Daily: Energy 700kcal, Protein 20g, 100% of recommended dietary allowance for all micronutrients during the 6 months of lactation. Vitamin A is excluded.
  Other Names: Produced by Nutriset. Daily dose: 2 sachets.
  Arms: Infant NVP & Nutrition Supplement; Maternal ARVs & Nutrition Supplement; No Drugs & Nutrition Supplement

SUMMARY:
This is a comparative clinical trial among HIV-infected women and their infants to determine:

1. the benefit of nutritional supplementation given to women during breastfeeding
2. the benefit and safety of antiretroviral (ARV) medications given either to infants or to their mothers to prevent HIV transmission during breastfeeding
3. the feasibility of exclusive breastfeeding followed by early, rapid breastfeeding cessation

DETAILED DESCRIPTION:
This study addresses the complex issues of HIV related maternal morbidity, mortality, and postnatal HIV transmission during breastfeeding and weaning in resource-poor countries. Objectives include assessment of mortality and morbidity among HIV-infected women; evaluation of interventions to reduce HIV transmission to infants exposed by breast milk; and assessment of early weaning as a risk-reduction strategy for infants of HIV-infected mothers.

The study will evaluate the following:

1. The efficacy of a high-density caloric/micronutrient nutritional supplement given to HIV-infected women who breastfeed in preventing maternal depletion (weight loss and micronutrient status).
2. The safety and efficacy of maternal or infant antiretroviral regimens, taken for up to 6 months during breastfeeding, in reducing infant HIV infection rates at 48 weeks.
3. The feasibility of exclusive breastfeeding for 6 months followed by rapid weaning.

Additional study objectives are to evaluate the feasibility of delivering these interventions in resource poor settings and to identify maternal, infant, and virologic factors associated with HIV transmission during breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

Recruitment and primary eligibility criteria:

* Age > 14 years.
* Ability to give informed assent or consent.
* Evidence of HIV infection, as documented by 2 positive ELISA antibody tests; or 1 positive ELISA, and 1 Western Blot; or 2 separate concurrent rapid tests.
* Currently pregnant (with a single or multiple fetuses).
* Gestation < 30 weeks at referral from 'Call to Action' Program
* No serious current complications of pregnancy.
* Intention to breastfeed.
* Intention to deliver at the institution at which the study is based.
* Not previously enrolled in this study for an earlier pregnancy.
* Other than HIV, no active serious infection, such as tuberculosis or other potentially serious illnesses.
* No previous use of antiretrovirals including the HIVNET 012 regimen.
* Mother's CD4 count > 250 cells/uL determined in the antenatal clinic.
* Mother's ALT < 2.5 x ULN (upper limit of normal) determined in the antenatal clinic

Secondary eligibility criteria and treatment assignment:

* Mother who delivers outside of the institution at which the study is based must present with her infant to the study site within 36 hours of delivery.
* Mother accepts nevirapine and zidovudine+lamivudine 7-day regimen for herself and her infant.
* Infant birth weight > 2000 g.
* No severe congenital malformations or other condition(s) not compatible with life.
* Based on clinical assessment, no maternal condition which would preclude the start of the study intervention.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2369 (Actual)
Dates: Start 2004-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Postpartum weight loss between delivery and 28 weeks | between delivery and 28 weeks
Infant HIV status at 28 weeks. (Infants found to have HIV at birth or 2 weeks after delivery will have been disenrolled.) | birth to 28 weeks
Exclusive breastfeeding and breastfeeding cessation by 28 weeks | birth to 28 weeks

SECONDARY OUTCOMES:
Duration of exclusive breastfeeding | birth to 28 weeks
Infant HIV status through 48 weeks | birth to 48 weeks
Maternal adherence to ARV, maternal CD4 count, and clinical assessment of opportunistic infection status through 48 weeks | delivery to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles van der Horst, MD, Study Chair — University of North Carolina, Chapel Hill; Denise J Jamieson, MD, MPH, Principal Investigator — CDC, Atlanta, GA; Peter Kazembe, MB ChB, Principal Investigator — Kamuzu Central Hospital
Locations (1):
- Kamuzu Central Hospital, Bottom Hospital, Lilongwe, Malawi

REFERENCES:
- [Derived] Flax VL, Adair LS, Allen LH, Shahab-Ferdows S, Hampel D, Chasela CS, Tegha G, Daza EJ, Corbett A, Davis NL, Kamwendo D, Kourtis AP, van der Horst CM, Jamieson DJ, Bentley ME; BAN Study Team. Plasma Micronutrient Concentrations Are Altered by Antiretroviral Therapy and Lipid-Based Nutrient Supplements in Lactating HIV-Infected Malawian Women. J Nutr. 2015 Aug;145(8):1950-7. doi: 10.3945/jn.115.212290. Epub 2015 Jul 8. PMID 26156797
- [Derived] Widen EM, Bentley ME, Chasela CS, Kayira D, Flax VL, Kourtis AP, Ellington SR, Kacheche Z, Tegha G, Jamieson DJ, van der Horst CM, Allen LH, Shahab-Ferdows S, Adair LS; BAN Study Team. Antiretroviral Treatment Is Associated With Iron Deficiency in HIV-Infected Malawian Women That Is Mitigated With Supplementation, but Is Not Associated With Infant Iron Deficiency During 24 Weeks of Exclusive Breastfeeding. J Acquir Immune Defic Syndr. 2015 Jul 1;69(3):319-28. doi: 10.1097/QAI.0000000000000588. PMID 25723140
- [Derived] Flax VL, Bentley ME, Combs GF Jr, Chasela CS, Kayira D, Tegha G, Kamwendo D, Daza EJ, Fokar A, Kourtis AP, Jamieson DJ, van der Horst CM, Adair LS. Plasma and breast-milk selenium in HIV-infected Malawian mothers are positively associated with infant selenium status but are not associated with maternal supplementation: results of the Breastfeeding, Antiretrovirals, and Nutrition study. Am J Clin Nutr. 2014 Apr;99(4):950-6. doi: 10.3945/ajcn.113.073833. Epub 2014 Feb 5. PMID 24500152
- [Derived] Widen EM, Bentley ME, Kayira D, Chasela CS, Daza EJ, Kacheche ZK, Tegha G, Jamieson DJ, Kourtis AP, van der Horst CM, Allen LH, Shahab-Ferdows S, Adair LS; BAN Study Team. Changes in soluble transferrin receptor and hemoglobin concentrations in Malawian mothers are associated with those values in their exclusively breastfed, HIV-exposed infants. J Nutr. 2014 Mar;144(3):367-74. doi: 10.3945/jn.113.177915. Epub 2013 Dec 31. PMID 24381222
- [Derived] Widen EM, Bentley ME, Kayira D, Chasela CS, Jamieson DJ, Tembo M, Soko A, Kourtis AP, Flax VL, Ellington SR, van der Horst CM, Adair LS; BAN Study team. Maternal weight loss during exclusive breastfeeding is associated with reduced weight and length gain in daughters of HIV-infected Malawian women. J Nutr. 2013 Jul;143(7):1168-75. doi: 10.3945/jn.112.171751. Epub 2013 May 22. PMID 23700341
- [Derived] Flax VL, Bentley ME, Chasela CS, Kayira D, Hudgens MG, Kacheche KZ, Chavula C, Kourtis AP, Jamieson DJ, van der Horst CM, Adair LS. Lipid-based nutrient supplements are feasible as a breastmilk replacement for HIV-exposed infants from 24 to 48 weeks of age. J Nutr. 2013 May;143(5):701-7. doi: 10.3945/jn.112.168245. Epub 2013 Mar 6. PMID 23468553
- [Derived] Flax VL, Bentley ME, Chasela CS, Kayira D, Hudgens MG, Knight RJ, Soko A, Jamieson DJ, van der Horst CM, Adair LS. Use of lipid-based nutrient supplements by HIV-infected Malawian women during lactation has no effect on infant growth from 0 to 24 weeks. J Nutr. 2012 Jul;142(7):1350-6. doi: 10.3945/jn.111.155598. Epub 2012 May 30. PMID 22649265
- [Derived] Jamieson DJ, Chasela CS, Hudgens MG, King CC, Kourtis AP, Kayira D, Hosseinipour MC, Kamwendo DD, Ellington SR, Wiener JB, Fiscus SA, Tegha G, Mofolo IA, Sichali DS, Adair LS, Knight RJ, Martinson F, Kacheche Z, Soko A, Hoffman I, van der Horst C; BAN study team. Maternal and infant antiretroviral regimens to prevent postnatal HIV-1 transmission: 48-week follow-up of the BAN randomised controlled trial. Lancet. 2012 Jun 30;379(9835):2449-2458. doi: 10.1016/S0140-6736(12)60321-3. Epub 2012 Apr 26. PMID 22541418
- [Derived] Chasela CS, Hudgens MG, Jamieson DJ, Kayira D, Hosseinipour MC, Kourtis AP, Martinson F, Tegha G, Knight RJ, Ahmed YI, Kamwendo DD, Hoffman IF, Ellington SR, Kacheche Z, Soko A, Wiener JB, Fiscus SA, Kazembe P, Mofolo IA, Chigwenembe M, Sichali DS, van der Horst CM; BAN Study Group. Maternal or infant antiretroviral drugs to reduce HIV-1 transmission. N Engl J Med. 2010 Jun 17;362(24):2271-81. doi: 10.1056/NEJMoa0911486. PMID 20554982